CLINICAL TRIAL: NCT04613700
Title: The Role of Secretin on the Energy Homeostasis
Acronym: THE-ROSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: The-ROSE
Record Dates: First submitted 2020-10-19; First posted 2020-11-03 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Obesity; Metabolic Disease; Diabetes; Adiposity
MeSH Terms: conditions — Obesity; Metabolic Diseases; Diabetes Mellitus | interventions — Secretin

STUDY DESIGN:
Intervention Model Description: randomised, double-blinded, placebo-controlled, cross-over study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secretin (Active Comparator)
  Interventions: Drug: Secretin
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Secretin — Native hormone
  Arms: Secretin
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
As of last year, new insight into the function of secretin was brought about as rodent studies showed secretin to possess potential body weight-regulating effects. In these studies, secretin was shown to increase non-shivering thermogenesis in brown adipose tissue (BAT), decrease meal size and promote meal discontinuation. The mechanisms behind these regulatory effect of secretin on energy homeostasis are unclear,

DETAILED DESCRIPTION:
Secretin was - as the first hormone - identified in 19021, but was not isolated until the 1960s. Secretin is produced in and secreted form small intestinal S cells. In the 1970s, the primary endocrine effects of secretin were unequivocally confirmed, namely potentiation of bicarbonate and pepsin secretion from the pancreas as well as stimulation of bile production in the liver. In the 1990s, the biosynthesis of secretin was delineated and its receptor was discovered. In the 2000s the pancreatic regulation of intestinal pH was shown to be secretin-mediated. As of last year, new insight into the function of secretin was brought about as rodent studies showed secretin to possess potential body weight-regulating effects. In these studies, secretin was shown to increase non-shivering thermogenesis in brown adipose tissue (BAT), decrease meal size and promote meal discontinuation.

The primary aim of this study is to evaluate the effect of a 5-hour intravenous infusion with the naturally occurring hormone secretin on ad libitum food intake (primary endpoint) compared to a double-blinded placebo (isotonic saline) infusion in 25 healthy young males.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Body mass index between 18.5 and 27.5 kg/m2
* Informed consent
* Body weight above 50 kg

Exclusion Criteria:

* Anaemia (blood haemoglobin below normal range)
* Known liver disease and/or alanine aminotransferase and/or aspartate transaminase > 2 times upper normal values
* Nephropathy (serum creatinine above normal range and/or albuminuria)
* Clinically significant kidney function impairment or other laboratory findings leading to the diagnosis of clinically relevant disorders (thyroid dysfunction, anaemia etc)
* Any physical or psychological condition that the investigators feel would interfere with trial participation

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Food intake on ad libitum meal | 300 minutes
  Kilojoule
Duration of ad libitum meal | 300 minutes
  Duration in minutes

SECONDARY OUTCOMES:
Water intake during ad libitum meal | 300 minutes
  mL
resting energy expenditure | Baseline, 90 minutes and 270 minutes
  Indirect calorimetry of respiration
Supraclavicular Brown adipose activity | -15 to 15 , 90 and 270 minutes
  Evaluated by neck skin temperature assessed using a non-invasive thermal imaging camera)
Appetite and satiety sensations (assessed by VASs), | Every 15 minutes after infusion, until time-point 90, hereafter every 30 minutes
  Visual analogue scales with a scale of 1-10 (Direction of scale varies)
Heart rate | every 15 minutes from from -15 to 300 minutes
  heart rate .
systolic blood pressure | every 15 minutes from from -15 to 300 minutes
  Systolic blood pressure
Diastolic blood pressure | every 15 minutes from from -15 to 300 minutes
  Diastolic blood pressures
Gallbladder motility | Timepoint -30, 10,20,45,60,75,90,120,210,300 minutes
  Gallbladder motility measured by Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, Professor, MD, Principal Investigator — Gentofte Hospital
Locations (1):
- Herlev- Gentofte Hospital, Center for Clinical Metabolic Research, Hellerup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heimburger SMN, Bentzen MJ, Kizilkaya HS, Hartmann B, Holst JJ, Rosenkilde MM, Dela F, Hansen SH, Rehfeld JF, Christensen MB, Knop FK. Secretin infusion decreases food intake in healthy men-a randomized, placebo-controlled, double-blind, crossover study. Eur J Endocrinol. 2024 Nov 27;191(6):545-557. doi: 10.1093/ejendo/lvae147. PMID 39556772